CLINICAL TRIAL: NCT05211973
Title: Developing Novel Digital Endpoints in Anorexia of Aging in Elderly Populations Residing in Long Term Care (LTC), Nursing Home, or Assisted Living Facilities
Brief Title: Geriatric Anorexia Study 2.0
Acronym: GAS2
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Other Study IDs: H-42048
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Healthy; Frailty
Keywords: Healthy; Wearable Devices; Geriatric Anorexia; Frail
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Fried Frailty Phenotype 0: Those who are considered Robust under the Fried Frailty Criteria. Sensor technology and digital measures will be used to evaluate movement and body weight composition in healthy adults.
  Interventions: Device: Wrist Actigraphy Device; Device: Smart Body Weight Scale; Device: Chair Scale; Device: Handheld Body Fat Percentage Device; Device: Bioelectric Impedance Analysis Scale
- Fried Frailty Phenotype 1-2: Those who are considered Intermediate/Pre-frail under the Fried Frailty Criteria. Sensor technology and digital measures will be used to evaluate movement and body weight composition in healthy adults.
  Interventions: Device: Wrist Actigraphy Device; Device: Smart Body Weight Scale; Device: Chair Scale; Device: Handheld Body Fat Percentage Device; Device: Bioelectric Impedance Analysis Scale
- Fried Frailty Phenotype 3+: Those who are considered Frail under the Fried Frailty Criteria. Sensor technology and digital measures will be used to evaluate movement and body weight composition in healthy adults.
  Interventions: Device: Wrist Actigraphy Device; Device: Smart Body Weight Scale; Device: Chair Scale; Device: Handheld Body Fat Percentage Device; Device: Bioelectric Impedance Analysis Scale

INTERVENTIONS:
Device: Wrist Actigraphy Device — a watch like wearable sensor
  Other Names: Geneactiv Watch
Device: Smart Body Weight Scale — a full body composition scale that provides fat and muscle mass, water retention, bone mass, and weight trends (conducted based on participant's abilities)
  Other Names: Renpho
Device: Chair Scale — a wheel-chair compatible scale to measure body weight
  Other Names: Meilestone
Device: Handheld Body Fat Percentage Device — a handheld device that measures body fat percentage
  Other Names: Omron
Device: Bioelectric Impedance Analysis Scale — a research-grade full body composition scale that provides fat and muscle mass, water retention, bone mass, and weight trends (conducted based on participant's abilities)
  Other Names: Tanita

SUMMARY:
Reduction in appetite and/or food intake among older individuals is referred to as anorexia of aging (AOA, also known as Geriatric Anorexia). AOA is linked with myriad comorbidities associated with aging, contributes significantly to adverse health consequences in old age, and has been used as a predictor of morbidity and mortality. The overall aim of this study is to compare feasibility of body weight, body fat, body composition and activity assessments in elderly subjects in long-term care (LTC), nursing home, or assisted living facilities. This will be accomplished through the use of questionnaires in addition to devices that evaluate movement, body composition, and body weight.

DETAILED DESCRIPTION:
The overall aim of this study is to compare feasibility of body weight, body fat, body composition and activity assessments in elderly subjects in long-term care (LTC), nursing home, or assisted living facilities. This will be accomplished through the use of questionnaires in addition to devices that evaluate movement, body composition, and body weight.

The proposed study will consist of an initial intake visit on Day 1, followed by an at-home (i.e. LTC facility, nursing home, and/or assisted living facility) phase where the participant will wear two watch like devices one on each wrist and answer two questions on paper each day. There will be a second visit on day 8 where the participant will complete additional questionnaires and assessments. The participant will continue wearing the wrist-worn devices for days 9-14, with a final visit on day 15 for final assessments and device collection. A window of +/- 3 days will be allocated for the scheduling of all visits to accommodate participant's schedules and commitments. Activities will take place in the care facility where the participant resides, or the Laboratory for Human Neurobiology for those that will commute. The study procedures will be identical for all participants for all Frailty groups.

ELIGIBILITY:
Inclusion Criteria: [separated into the three groups based on the Fried Criteria: 0 - robust, 1-2 - intermediate or pre-frail, 3 or above - frail; enrollment into individual frailty groups will close once the recruitment goal is reached for that group]

1. Male or female participants aged 65 years of age and over
2. No recent hospitalizations/acute events in last 30 days
3. No active or recent (within 12 months) cancer diagnosis except skin cancer [limited to only non-complicated squamous and basal cell skin cancer (SCC/BCC)]
4. Body mass index (BMI) < 30 kg/m2
5. Able to understand and cooperate with study procedures and able to read, understand and provide informed consent. Evidence of a personally signed and dated informed consent document indicating that the participant, if necessary, their legally authorized representative (LAR) has been informed of all pertinent aspects of the study.
6. Native English speakers or demonstrated fluency in English as determined by the Investigator
7. WRAT-4 Word Reading Subtest equivalent to 8th grade reading level or greater
8. Montreal Cognitive Assessment (MoCA) score of ≥ to 19

Exclusion Criteria:

1. Treatment with an investigational drug within 30 days of enrollment
2. Moderate to severe alcohol use disorder diagnosis within 6 months of the screening as disclosed by the subject
3. Participants who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or participants who are Boston University/Boston Medical Center (BU/BMC) employees directly involved in the conduct of the study
4. Inability to comply with study requirements
5. Life expectancy of less than 6 months, or actively enrolled in a palliative care program
6. Has any clinically significant medical disorder, condition, disease, or clinically significant finding at screening that precludes subject's participation in study activities
7. Participants with electronic implant such as pacemaker etc., due to Bioelectric Impedance Analysis (BIA) body composition devices (Tanita, Smart body scale) using tiny electrical signal for measurements
8. At an increased risk of COVID-19 as determined by the Laboratory for Human Neurobiology COVID-19 Human Subject Risk Assessment Survey
9. Temperature equal to or above 100.4 degrees F
10. Modified Barthel Index of <40

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Healthy Adults
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Assess the use of accelerometry in an elderly cohort based in a LTC/nursing home/assisted-living setting | 2 weeks +/- 3 days
  Two GENEActiv watches will be used (one on each wrist) at a sampling rate of 50 Hz to measure movement in the x, y, and z direction across the study period.
Assess the use of a smart standing scale for body weight and composition assessment in an elderly cohort based in a LTC/nursing home/assisted-living setting (based on participant's abilities). | 2 weeks +/- 3 days
  A body weight composition scale will be used to completion of daily weight measurement and track body weight in kilograms (kg) throughout the study (based on participant's abilities).
Assess the use of a chair scale for body weight assessment in an elderly cohort based in a LTC/nursing home/assisted-living setting. | 2 weeks +/- 3 days
  A chair scale will be used during study staff visits to measure and track body weight.
Assess the use of a handheld body fat assessment tool for body fat percentage assessment in an elderly cohort based in a LTC/nursing home/assisted-living setting. | 2 weeks +/- 3 days
  A handheld body fat assessment tool will be used during study staff visits to measure body fat percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Thomas, PhD, MBA, Principal Investigator — Principal Investigator, Boston University, Department of Anatomy & Neurobiology
Locations (1):
- Evans Biomedical Research Center, Boston, Massachusetts, United States